CLINICAL TRIAL: NCT01820273
Title: Study of Incretins Response and Glycemic Control: Pre Diet, After Conventional Weight Loss and in the Early Postoperative Phase After Gastric Bypass in T2D-patients.
Brief Title: Changes in Incretins Response and Glycemic Control After Gastric Bypass Surgery in Type 2 Diabetic Patients Versus Healthy
Status: Withdrawn | Type: Observational
Why Stopped: Study no longer at LU.
Sponsor: Lund University (Other)
Collaborators: Kalmar County Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: MRD-Study
Record Dates: First submitted 2013-03-25; First posted 2013-03-28 (Estimated); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Type 2 Diabetes; Obesity
Keywords: Type 2 diabetes; Bariatric surgery; incretines; GLP-1; GIP; gastric bypass; foregut; hindgut
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Bloodsamples
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine the early changes in gut hormonal, and other metabolites with known relations to the glycemic homeostasis. The study mainly focus on these responses to food in the diabetic patient, compared to the non-diabetic, after gastric bypass surgery. Also aiming for recording changes in the earliest postoperative phase.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of type 2 diabetes
* obesity BMI >35

Exclusion Criteria:

* prior bariatric surgery

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: female obese (BMI>35)patients accepted for bariatric surgery (lap gastric bypass). 10 patients with type 2 diabetes(T2D) 6 10 matched controls without T2D.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2013-04; Primary Completion 2016-05-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
changes in incretines in the bariatric patient | 2 months prior to surgery - 6 weeks post surgery
  standardized meals prior to pre op diet, day before surgery, first day after surgery and 6 weeks after surgery.

SECONDARY OUTCOMES:
Diabetes control | 6 weeks post surgery
  resolution of t2D as early as first day after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Nils Wierup, Study Director — Lunds Universitet, Clinical researchcenter; Johan Berggren, MD, Principal Investigator — Lunds Universitet
Locations (1):
- Kalmar County Hospital, Kalmar, Sweden